CLINICAL TRIAL: NCT02188784
Title: Oral Iron Repletion Effects On Oxygen Uptake in Heart Failure
Acronym: IRONOUT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Adrian Hernandez (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, Adrian Hernandez, MD, MHS, FAHA: Associate Professor of Medicine;Director, Outcomes & Health Services Research, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00054061; 2U10HL084904 (NIH)
Record Dates: First submitted 2014-07-10; First posted 2014-07-14 (Estimated); Results first posted 2017-05-15 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-06

CONDITIONS: Chronic Heart Failure
MeSH Terms: interventions — Niferex

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Polysaccharide iron complex 150 mg (Active Comparator): oral Fe polysaccharide 150mg twice daily for 16 weeks
  Interventions: Drug: Polysaccharide Iron Complex 150 mg
- Placebo (for Polysaccharide Iron Complex 150 mg) (Placebo Comparator): Oral placebo twice a day for 16 weeks
  Interventions: Drug: Placebo (for Polysaccharide Iron Complex)

INTERVENTIONS:
Drug: Polysaccharide Iron Complex 150 mg — Oral Iron
  Other Names: Feramax 150 mg
  Arms: Polysaccharide iron complex 150 mg
Drug: Placebo (for Polysaccharide Iron Complex) — Sugar capsule designed to mimic Polysaccharide Iron Complex.
  Arms: Placebo (for Polysaccharide Iron Complex 150 mg)

SUMMARY:
The purpose of this study is to determine if oral iron (Fe) polysaccharide is superior to oral placebo in improving functional capacity as measured by change in peak VO2 (oxygen uptake) by CPET (Cardiopulmonary Exercise Testing) , of a broad population of patients with HFrEF (Heart Failure with Reduced Ejection Fraction) and Fe deficiency at 16 weeks.

Hypothesis: In a broad population of HFrEF patients with Fe deficiency, compared to oral placebo, therapy with oral Fe polysaccharide will be associated with improvement in functional capacity at 16 weeks as assessed by CPET.

DETAILED DESCRIPTION:
Therapeutic options to further improve functional capacity and symptoms in HF beyond neurohormonal antagonism are limited. Studies have demonstrated impaired oxidative capacity of skeletal muscle among HF patients, which may contribute to symptoms of breathlessness and persistent fatigue.

In addition to its role in erythropoiesis, iron (Fe) plays a critical role in skeletal muscle's oxygen (O2)-storage capacity (myoglobin) and systemic aerobic energy production. As Fe deficiency is common in patients with symptomatic HF, repletion of iron stores may improve submaximal exercise capacity among these patients beyond the effects on erythropoiesis.

While intravenous Fe repletion in HF patients with mild Fe-deficiency (i.e. Ferritin <100 or Ferritin 100-299 with transferrin saturation <20%) with or without anemia global well-being and functional status, oral Fe repletion has not been studied. Furthermore, the efficacy of oral Fe to replete iron stores in a similar population and its impact on functional capacity, measured objectively by peak VO2, remains unknown.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years
2. Previous clinical diagnosis of heart failure with current New York Heart Association (NYHA) Class II-IV symptoms LVEF≤0.40 within 2 years prior to consent, and ≥3 months after a major change in cardiac status (i.e. CABG or CRT).
3. Serum ferritin between 15-100 ng/ml or serum ferritin between 100-299 ng/ml with transferrin saturation <20%
4. Hemoglobin 9.0-13.5 g/dL (males), 9-13.5 (females) at time of enrollment
5. Stable evidence-based medical therapy for HF (including beta-blocker and ACE-inhibitor/ARB unless previously deemed intolerant, and diuretics as necessary) with </= 100% change in dose for 30 days prior to randomization

   a. Changes in diuretic dose guided by a patient-directed flexible dosing program are considered stable medical therapy
6. Willingness to provide informed consent

Exclusion Criteria:

1. Presence of a neuromuscular, orthopedic or other non-cardiac condition that prevents the patient from exercise testing on a bicycle/treadmill ergometer and/or inability to achieve an RER ≥ 1.0 on screening/baseline CPET
2. Severe renal dysfunction (eGFR< 20 ml/min/1.73m2)
3. Severe liver disease (ALT or AST > 3x normal, alkaline phosphatase or bilirubin >2x normal)
4. Gastrointestinal conditions known to impair Fe absorption (i.e. inflammatory bowel disease)
5. Known active infection as defined by current use of oral or intravenous antimicrobial agents
6. Documented active gastrointestinal bleeding
7. Active malignancy other than non-melanoma skin cancers
8. Anemia with known cause other than Fe deficiency or chronic disease
9. Fe overload disorders (i.e. hemochromatosis or hemosiderosis)
10. History of erythropoietin, IV or oral Fe therapy, or blood transfusion in previous 3 months.
11. Current ventricular assist device
12. Anticipated cardiac transplantation within the next 4 months
13. Primary hypertrophic cardiomyopathy, infiltrative cardiomyopathy, acute myocarditis, constrictive pericarditis or tamponade
14. Previous adverse reaction to study drug or other oral Fe preparation
15. Known or anticipated pregnancy in the next 4 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2014-09-03 (Actual); Primary Completion 2016-04-06 (Actual); Study Completion 2016-04-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Hernandez, MD,MHS,FAHA, Principal Investigator — Duke University
Locations (17):
- United States (17):
  - Emory University School of Medicine, Atlanta, Georgia
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Saint Louis University Hospital, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Duke University Medical Center, Durham, North Carolina
  - University Hospitals-Case Medical Center, Cleveland, Ohio
  - Metor Health System, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Utah Hospitals and Clinics, Murray, Utah
  - The University of Vermont - Fletcher Allen Health Care, Burlington, Vermont

IPD SHARING:
Plan to Share IPD: Yes
After the study results have been published, site-specific participant data will be shared with sites upon request. Sites are expected to follow their specific institutional policies regarding sharing results with their participants.

REFERENCES:
- [Derived] Lewis GD, Malhotra R, Hernandez AF, McNulty SE, Smith A, Felker GM, Tang WHW, LaRue SJ, Redfield MM, Semigran MJ, Givertz MM, Van Buren P, Whellan D, Anstrom KJ, Shah MR, Desvigne-Nickens P, Butler J, Braunwald E; NHLBI Heart Failure Clinical Research Network. Effect of Oral Iron Repletion on Exercise Capacity in Patients With Heart Failure With Reduced Ejection Fraction and Iron Deficiency: The IRONOUT HF Randomized Clinical Trial. JAMA. 2017 May 16;317(19):1958-1966. doi: 10.1001/jama.2017.5427. PMID 28510680
- [Derived] Lewis GD, Semigran MJ, Givertz MM, Malhotra R, Anstrom KJ, Hernandez AF, Shah MR, Braunwald E. Oral Iron Therapy for Heart Failure With Reduced Ejection Fraction: Design and Rationale for Oral Iron Repletion Effects on Oxygen Uptake in Heart Failure. Circ Heart Fail. 2016 May;9(5):e000345. doi: 10.1161/CIRCHEARTFAILURE.115.000345. PMID 27140203

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Polysaccharide Iron Complex 150 mg | Placebo (for Polysaccharide Iron Complex 150 mg)
Started | 111 | 114
Completed | 102 (Patients completing the protocol excluding death, lost to follow-up and withdrawn consent.) | 101 (Patients completing the protocol excluding death, lost to follow-up and withdrawn consent.)
Not Completed | 9 | 13
Not completed — Death | 3 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 3 | 9
Not completed — Physician Decision | 2 | 3

BASELINE CHARACTERISTICS:
Population: All randomized patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Polysaccharide Iron Complex 150 mg | Placebo (for Polysaccharide Iron Complex 150 mg) | Total
Number analyzed (Participants) | 111 | 114 | 225
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.8 (13.4) | 51.6 (12.5) | 61.7 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 36 | 80
  Male | 67 | 78 | 145
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 6 | 9
  Not Hispanic or Latino | 108 | 107 | 215
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 31 | 26 | 57
  White | 79 | 85 | 164
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 111 | 114 | 225

OUTCOME MEASURES:

1. Primary Outcome: Change in Peak VO2 (ml/Min) (VO2 =Oxygen Consumption)
Description: To determine if oral Fe (Iron) polysaccharide is superior to oral placebo in improving functional capacity as measured by change in peak VO2 by CPET (Cardiopulmonary Exercise Testing) , of a broad population of patients with HFrEF (Heart Failure with Reduced Ejection Fraction) and Fe deficiency at 16 weeks.
Time Frame: Baseline (BL) and Week 16
Population: All randomized patients with available change data
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Polysaccharide Iron Complex 150 mg | Placebo (for Polysaccharide Iron Complex 150 mg)
Number analyzed (Participants) | 96 | 95
mL/min | 28.04 (212.75) | 3.90 (190.24)
Statistical Analysis 1: Comparison: Polysaccharide Iron Complex 150 mg vs Placebo (for Polysaccharide Iron Complex 150 mg); Test type: Superiority or Other; p = 0.4570, Regression, Linear; Mean Difference (Net) = 21.03, 95% CI 2-sided [-34.38 to 76.43]

2. Secondary Outcome: Change From Baseline in Sub-maximal Exercise Capacity as Assessed by the 6 Minute Walk Test (6MWT)
Description: To determine the impact of oral Fe repletion on Submaximal exercise capacity as measured by 6MWT
Time Frame: Measured at BL, week 8 and week 16
Population: All randomized patients with available change data
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Polysaccharide Iron Complex 150 mg | Placebo (for Polysaccharide Iron Complex 150 mg)
Number analyzed (Participants) | 111 | 114
meters
  8 weeks: number analyzed (Participants) | 101 | 97
  8 weeks | 12.65 (95.89) | 16.63 (83.20)
  16 weeks: number analyzed (Participants) | 97 | 97
  16 weeks | 10.76 (62.29) | 30.94 (77.33)
Statistical Analysis 1: Comparison: Polysaccharide Iron Complex 150 mg vs Placebo (for Polysaccharide Iron Complex 150 mg); Change from Baseline to Week 8; Test type: Superiority or Other; p = 0.9487, Regression, Linear; Mean Difference (Net) = -0.77, 95% CI 2-sided [-24.12 to 22.59]
Statistical Analysis 2: Comparison: Polysaccharide Iron Complex 150 mg vs Placebo (for Polysaccharide Iron Complex 150 mg); Change from Baseline to Week 16; Test type: Superiority or Other; p = 0.1921, Regression, Linear; Mean Difference (Net) = -12.67, 95% CI 2-sided [-31.71 to 6.37]

3. Secondary Outcome: Change in Plasma NT-pro BNP
Description: To determine the impact of oral Fe repletion on Plasma N-terminal pro-B-type natriuretic peptide (NT-pro BNP)
Time Frame: Measured at Baseline and Week 16
Population: All randomized patients with available change data
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Polysaccharide Iron Complex 150 mg | Placebo (for Polysaccharide Iron Complex 150 mg)
Number analyzed (Participants) | 98 | 98
pg/ml | 119.36 (1937.58) | -70.88 (1256.49)
Statistical Analysis 1: Comparison: Polysaccharide Iron Complex 150 mg vs Placebo (for Polysaccharide Iron Complex 150 mg); Test type: Superiority or Other; p = 0.4296, Regression, Linear; Mean Difference (Net) = 182.43, 95% CI 2-sided [-272.14 to 637.0]

4. Secondary Outcome: Change in Health Status: Kansas City Cardiomyopathy Questionnaire (KCCQ) - Clinical Summary Score
Description: To determine the impact of oral Fe repletion on Health Status: KCCQ.
  KCCQ is a 23-item, self administered instrument that quantifies physical function, symptoms (frequency, severity and recent change), social function, self-efficacy and knowledge, and quality of life for patients with congestive heart failure. It is a predictive tool that tracks how patients are doing if they have weakened heart muscle due to prior heart attacks, heart valve problems, viral infections, or other causes.
  The KCCQs questions are used to calculate scores in ten domains. Physical Limitation, Symptom Stability, Frequency, Burden and Total Symptom. Social Limitation, Self-Efficacy, Quality of Life, and Clinical Summary. Overall summary: a combined measure of all the above.
  For each domain, the validity, reproducibility, responsiveness and interpretability have been independently established. Scores are transformed to a range of 0-100, in which higher scores reflect better health status.
Time Frame: Measured at Baseline, Week 8 and Week 16
Population: All randomized patients with available change data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Polysaccharide Iron Complex 150 mg | Placebo (for Polysaccharide Iron Complex 150 mg)
Number analyzed (Participants) | 111 | 114
units on a scale
  Week 8: number analyzed (Participants) | 104 | 103
  Week 8 | 3.25 (16.91) | 0.58 (13.63)
  Week 16: number analyzed (Participants) | 100 | 100
  Week 16 | 3.42 (16.05) | 4.11 (11.80)
Statistical Analysis 1: Comparison: Polysaccharide Iron Complex 150 mg vs Placebo (for Polysaccharide Iron Complex 150 mg); Change from baseline to week 8; Test type: Superiority or Other; p = 0.0722, Regression, Linear; Mean Difference (Net) = 3.60, 95% CI 2-sided [-0.33 to 7.52]
Statistical Analysis 2: Comparison: Polysaccharide Iron Complex 150 mg vs Placebo (for Polysaccharide Iron Complex 150 mg); Change from baseline to week 16; Test type: Superiority or Other; p = 0.6927, Regression, Linear; Mean Difference (Net) = 0.71, 95% CI 2-sided [-2.83 to 4.24]

5. Secondary Outcome: Change From Baseline in O2 Uptake Kinetics as Assessed by Mean Response Time From CPET
Description: To determine the impact of oral Fe repletion on O2 Uptake Kinetics as measured by CPET
Time Frame: Measured at BL week 16
Population: All randomized patients with available change data
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Polysaccharide Iron Complex 150 mg | Placebo (for Polysaccharide Iron Complex 150 mg)
Number analyzed (Participants) | 71 | 62
seconds | 2.63 (13.31) | -0.95 (13.29)
Statistical Analysis 1: Comparison: Polysaccharide Iron Complex 150 mg vs Placebo (for Polysaccharide Iron Complex 150 mg); Test type: Superiority or Other; p = 0.0643, Regression, Linear; Mean Difference (Net) = 3.56, 95% CI 2-sided [-0.21 to 7.33]

6. Secondary Outcome: Change From Baseline in Ventilatory Efficiency Defined by Ve/VCO2
Description: Change from baseline in Ventilatory Efficiency defined by Ve/VCO2 (carbon dioxide output) as measured by CPET
Time Frame: Measured at BL week 16
Population: All randomized patients with available change data
Measure: Mean (Standard Deviation); unit: VE/VCO2 Slope
Arm/Group | Polysaccharide Iron Complex 150 mg | Placebo (for Polysaccharide Iron Complex 150 mg)
Number analyzed (Participants) | 96 | 95
VE/VCO2 Slope | -0.48 (5.85) | -1.31 (8.85)
Statistical Analysis 1: Comparison: Polysaccharide Iron Complex 150 mg vs Placebo (for Polysaccharide Iron Complex 150 mg); Test type: Superiority or Other; p = 0.4006, Regression, Linear; Mean Difference (Net) = 0.77, 95% CI 2-sided [-1.04 to 2.58]

ADVERSE EVENTS:
Time Frame: Randomization to Week 16
Arm/Group | Polysaccharide Iron Complex 150 mg | Placebo (for Polysaccharide Iron Complex 150 mg)
Serious Adverse Events (participants affected / at risk) | 11/111 | 9/114
Other Adverse Events (participants affected / at risk) | 18/111 | 24/114
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Polysaccharide Iron Complex 150 mg (N=111) | Placebo (for Polysaccharide Iron Complex 150 mg) (N=114)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Non-Cardiac Chest Pain (General disorders) | 2 (2) | 0 (0)
Bronchitis Viral (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis Viral (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 4 (4) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Streptococcal Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Vestibular Neuronitis (Infections and infestations) | 0 (0) | 1 (1)
Abdominal Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Liver Function Test Abnormal (Investigations) | 0 (0) | 1 (1)
Norovirus Test Positive (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hyperosmolar Hyperglycaemic State (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Skin Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Alcohol Withdrawal Syndrome (Psychiatric disorders) | 0 (0) | 1 (1)
Hypertensive Crisis (Vascular disorders) | 1 (1) | 0 (0)
Temporal Arteritis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Polysaccharide Iron Complex 150 mg (N=111) | Placebo (for Polysaccharide Iron Complex 150 mg) (N=114)
Abdominal Discomfort (Gastrointestinal disorders) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 6 (8) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 7 (7) | 4 (4)
Nausea (Gastrointestinal disorders) | 1 (1) | 4 (4)
Asthenia (General disorders) | 1 (1) | 2 (2)
Non-Cardiac Chest Pain (General disorders) | 0 (0) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Gout (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 2 (2) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
To minimize the probability of inaccurate data in published materials, it is the policy of The Heart Failure Network (HFN) that all data and text considered for all papers, and all abstracts for presentation at scientific meetings, be submitted to the Publication & Presentation Subcommittee, the NHLBI Project Officer and the Coordinating Center for review and approval prior to presentation or publication.